CLINICAL TRIAL: NCT02213783
Title: Comparison of the Pharmacodynamics of Imipenem in Patients With Febrile Neutropenia Following Administration by 4-hour Infusion and Bolus Injection.
Brief Title: Comparison of the Pharmacodynamics of Imipenem in Patients With Febrile Neutropenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMIFN53-068-11-1-1
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Patients With Febrile Neutropenia
Keywords: Imipenem; Febrile neutropenia; Gram-negative infection; Pharmacodynamic; Monte Carlo Simulation
MeSH Terms: conditions — Febrile Neutropenia | interventions — Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional arm (Active Comparator): Infusion of 0.5 g of imipenem for 0.5 hr every 6 hr for 2-5 days
  Interventions: Drug: Imipenem
- Extended infusion arm (Experimental): Infusion of 0.5 g of imipenem for 4 hr every 6 hr for 2-5 days
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Imipenem — Each patient will receive 0.5 g of imipenem, 0.5 hr infusion every 6 hr at room temperature
  Other Names: Tienam
  Arms: Conventional arm
Drug: Imipenem — Each patient will receive 0.5 g of imipenem, 4 hr infusion every 6 hr of at room temperature
  Other Names: Tienam
  Arms: Extended infusion arm

SUMMARY:
This is prospective and randomized study to compare the pharmacodynamics (t>MIC) of 0.5 g every 6 h of imipenem in twelve patients with febrile neutropenia following administration by a 4 h infusion or bolus injection.

Concentration of imipenem in plasma will be measured by HPLC method and simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to %PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > or = 20 years
* Patients who have febrile neutropenia with Gram negative bacilli infections which are sensitive to imipenem by the disk diffusion
* Patients who are likely to survive 3 days

Exclusion Criteria:

* Patients who have documented hypersensitivity to imipenem or other carbapenems
* Patients who have an estimated creatinine clearance of < 50 ml/min
* Patients who are in circulatory shock or hypotension (systolic < 90 mmHg)
* Patients who are pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Concentration of imipenem in plasma | 6 hours profile after 8th dose of imipenem
  Concentration of imipenem in plasma will be determined by HPLC method and simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response).

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, M.D., Principal Investigator — Prince of Songkla University
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand